CLINICAL TRIAL: NCT07103356
Title: Developing a Hybrid Type 1 Effectiveness-Implementation Randomized Controlled Trial to Test a Table-Top Water Pitcher to Reduce Arsenic Exposure in Northern New England
Brief Title: Table-Top Water Pitcher to Reduce Arsenic Exposure Among Well Users in New Hampshire
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Caitlin G. Howe, Assistant Professor of Epidemiology, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00033185
Record Dates: First submitted 2025-05-08; First posted 2025-08-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Arsenic Poisoning; Environmental Exposure; Water-Related Diseases
Keywords: Arsenic; Private Well; Environmental Health; Filter
MeSH Terms: conditions — Arsenic Poisoning; Waterborne Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Water Pitcher Filtration System (Experimental): Arm 1: No reminders to change water pitcher filter cartridges Arm 2: Weekly reminders to change water pitcher filter cartridges
  Interventions: Behavioral: Water Pitcher Filtration System

INTERVENTIONS:
Behavioral: Water Pitcher Filtration System — Table-top water pitcher filtration system

SUMMARY:
The goals of this clinical trial are to:

1. gather preliminary data on the effectiveness of a table-top water pitcher filtration system in reducing arsenic exposure among individuals using private wells with elevated (>5 μg/L) arsenic concentrations, and
2. identify the factors influencing implementation of the filter intervention (uptake and sustainability) and barriers and facilitators to its use.

The main questions it aims to answer are:

Do water and urinary arsenic concentrations change from baseline to Week 4 of the water pitcher intervention?

Are changes in arsenic concentrations maintained during the eight-week sustainability period?

* Which factors facilitate or impede uptake, use, and sustainability of the intervention?
* Are household income and/or home ownership associated with sustained filter use?

Participants will:

* Receive a free 12-cup water filter pitcher and cartridge replacements
* Use the pitcher filtration system, including replacement of filter cartridges, per manufacturer recommendations
* Collect and mail water and urine samples at baseline, 4 weeks, and 12 weeks
* Complete online questionnaires at baseline, 4 weeks, and 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* NH resident
* Receiving primary care at Dartmouth Hitchcock Clinics - Concord
* Use a private water system as primary drinking water source
* Do majority (>50%) of food preparation in home
* Interested in receiving a free water arsenic test kit
* Water arsenic >5 micrograms/L upon testing

Exclusion Criteria:

* Use or plan to use a mitigation strategy to reduce exposure to arsenic-contaminated drinking water

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Water arsenic concentrations | 4 weeks
  Changes in water arsenic concentrations from baseline to week 4
Urinary arsenic concentrations | 4 weeks
  Changes in urinary arsenic concentrations from baseline to week 4
Reach | 4 weeks
  Number of participants who receive the water pitcher filtration system among all eligible individuals and demographics
Adoption | 4 weeks
  Number of participants using the filtration system after receiving it; number of participants who intend to use the system after the study period ends; and demographics of participants who used the filtration system during the study period or intend to use it after the study period ends
Implementation | 4 weeks
  % of participants who adhere to the intervention during the intervention period (Fidelity), including using the pitcher filtration system for all drinking and cooking water and changing filter cartridges as recommended (measured by questionnaire: at home, did you use the pitcher filtration system for all of your drinking water, more than half of your drinking water, half of your drinking water, less than half of your drinking water, or none of your drinking water AND did you use did you use the pitcher filtration system for all of your cooking water, more than half of your cooking water, half of your cooking water, less than half of your cooking water, or none of your cooking water)
Maintenance | 8 weeks
  % of participants who continue to use the pitcher filtration system during the 8-week sustainability period when replacement filter cartridges are no longer provided (measured by questionnaire: at home, did you use the pitcher filtration system for all of your drinking water, more than half of your drinking water, half of your drinking water, less than half of your drinking water, or none of your drinking water AND did you use did you use the pitcher filtration system for all of your cooking water, more than half of your cooking water, half of your cooking water, less than half of your cooking water, or none of your cooking water)